CLINICAL TRIAL: NCT02516137
Title: Clinical Effects of Dry Needling Among Asymptomatic Individuals With Hamstring Tightness
Brief Title: Hamstring Tightness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Marie Johanson, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00077095
Record Dates: First submitted 2015-08-03; First posted 2015-08-05 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Hamstring Tightness
Keywords: Dry needling
MeSH Terms: interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dry needling group (Experimental): Subjects with tight hamstrings will receive dry needling to the hamstrings with the needle inserted into the muscle tissue in addition to a standard hamstring stretching exercise program.
  Interventions: Procedure: Dry needling; Other: Standard hamstring stretching exercise
- Sham dry needling group (Sham Comparator): Subjects with tight hamstrings will receive sham dry needling to the hamstrings with the needle inserted into the subcutaneous tissue in addition to a standard hamstring stretching exercise program.
  Interventions: Procedure: Sham needling; Other: Standard hamstring stretching exercise
- No needling group (Placebo Comparator): Subjects with tight hamstrings will receive no needling but have the tip of a blunt needle handle placed on the skin over the hamstrings in addition to a standard hamstring stretching exercise program.
  Interventions: Procedure: Blunt needle placement; Other: Standard hamstring stretching exercise

INTERVENTIONS:
Procedure: Dry needling — Dry needling will be performed on two points over the hamstring muscles on the randomly determined side. Points 2 cm distal to the ischial tuberosity and halfway between the ischial tuberosity and popliteal crease within the medial and lateral muscle bellies will be identified and the skin cleansed with rubbing alcohol. A Seirin L- type 50 mm needle will be inserted into each of the two points to a depth no greater than three-quarters length of the needle into the hamstring muscle for 30 seconds using a vertical pistoning technique and then statically up to 10 minutes.
  Arms: Dry needling group
Procedure: Sham needling — Sham dry needling will be performed on two points over the hamstring muscles on the randomly determined side. Points 2 cm distal to the ischial tuberosity and halfway between the ischial tuberosity and popliteal crease within the medial and lateral muscle bellies will be identified and the skin cleansed with rubbing alcohol. The plastic tube of a Seirin L- type 50 mm needle will be placed against the skin and the needle will be tapped once so that it is inserted subcutaneously no deeper than 5 mm for 30 seconds using a vertical pistoning technique and then statically up to 10 minutes in each location.
  Arms: Sham dry needling group
Procedure: Blunt needle placement — Blunt needle placement will be performed on two points over the hamstring muscles on the randomly determined side. Points 2 cm distal to the ischial tuberosity and halfway between the ischial tuberosity and popliteal crease within the medial and lateral muscle bellies will be identified and the skin cleansed with rubbing alcohol. A blunt needle handle is inserted into a plastic tube which will be placed over the identified points for 30 seconds and then for an additional 10 minutes each. The blunt needle handle only touches the skin without puncturing it.
  Arms: No needling group
Other: Standard hamstring stretching exercise — Subjects will be instructed to stretch the back of their thighs, once a day for 3 repetitions, holding for 30 seconds each time performed bilaterally.

SUMMARY:
The purpose of this study is to find out if individuals with tight hamstring muscles who receive dry needling in addition to a standard stretching exercise program, show an improvement in hamstring tightness and function compared to individuals with tight hamstrings who receive either sham dry needling or no needling (blunt needle) in addition to a standard stretching program.

DETAILED DESCRIPTION:
Tightness of the hamstring muscles is a risk factor for injury. Currently, there is no data on the effect of dry needling on hamstring extensibility or functional performance measures among asymptomatic individuals with hamstring muscle tightness. The investigator wants to assess if individuals with tight hamstring muscles who receive dry needling in addition to a standard stretching exercise program, exhibit reduced hamstring tightness and improved functional performance compared to individuals with tight hamstrings who receive either sham dry needling or no needling (blunt needle) in addition to a standard stretching program.

ELIGIBILITY:
Inclusion Criteria:

* Hamstring 90/90 extensibility goniometric measurement of more than 20 degrees of knee flexion bilaterally
* Ability to perform a squat to 90 degrees of knee flexion without assistance of the upper extremities
* Asymptomatic during walking

Exclusion Criteria:

* History of systemic neurological or arthritic condition
* History of bony or peripheral nerve trauma or surgery lower extremities
* History of treatment with dry needling
* No contraindications to dry needling

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-07; Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Change in hamstring muscle extensibility | Baseline, at 5 weeks from baseline
  Bilateral 90/90 hamstring muscle extensibility passive range of motion (PROM) measurements will be assessed using a goniometer. The goniometer measures the angle of the joint at both extremes of the range of motion (ROM). An increase in the passive range of motion (PROM) indicates increased hamstring muscle extensibility.
Change in unilateral hop for distance test scores | Baseline, at 5 weeks from baseline
  The functional performance of the hamstring muscles will be assessed by using the unilateral hop for distance test. The subjects will be instructed to stand on the leg to be tested and hop and land on the same limb. The distance hopped, measured at the level of the great toe, will be measured (centimeters). Scores will be recorded as absolute distance (in centimeters). An increase in the score (distance covered) from baseline to 5 weeks from baseline indicates better functional performance of the hamstrings.
Change in crossover hop for distance tests scores | Baseline, at 5 weeks from baseline
  The functional performance of the hamstring muscles will be assessed by using the crossover hop for distance test. The subjects will be instructed to hop forward 3 times while alternately crossing over a marking. The total distance hopped forward will be recorded. The heel of the hop leg will be used to determine the length of the jump. Crossover hop limb symmetry index (LSI) scores for knee function within normal ranges are generally greater than 95%. An increase in the crossover hop limb symmetry index (LSI) from baseline to 5 weeks from baseline indicates better functional performance of the hamstrings.

SECONDARY OUTCOMES:
Change in dynamometry pressure readings | Baseline, at 5 weeks from baseline
  The strength of the hamstrings will be assessed using a hand-held dynamometer.The subjects will be asked to exert maximal force against the dynamometer and the reading is recorded. Scores are based on force production in kilograms or pounds; kilograms (0-90), pounds (0-200). Higher pressure scores indicate better muscle strength of the hamstring muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Johanson, PT, PhD, OCS, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory Clinic, Atlanta, Georgia
  - Emory University, Atlanta, Georgia